CLINICAL TRIAL: NCT01475058
Title: A Phase I/II Study of Cellular Immunotherapy With Donor Central Memory-derived Virus-specific CD8+ T-cells Engineered to Target CD19 for CD19+ Malignancies After Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: CD19 CAR T Cells for B Cell Malignancies After Allogeneic Transplant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Cameron Turtle, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2494.00; NCI-2011-01819 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2494.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); R01CA136551 (NIH)
Record Dates: First submitted 2011-11-10; First posted 2011-11-21 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Philadelphia Chromosome Negative Adult Precursor Acute Lymphoblastic Leukemia; Philadelphia Chromosome Positive Adult Precursor Acute Lymphoblastic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Mantle Cell Lymphoma; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (T cell therapy) (Experimental): Patients undergo one IV infusion of donor-derived CD8+ central memory-derived CMV/CD19 or EBV/CD19 bi-specific T cells, at least 30 days after HCT.
  Interventions: Biological: allogeneic cytomegalovirus-specific cytotoxic T lymphocytes

INTERVENTIONS:
Biological: allogeneic cytomegalovirus-specific cytotoxic T lymphocytes — Allogeneic CD19-specific chimeric antigen receptor-modified CD8+ central memory derived virus-specific T cells. Allogeneic CD19CAR-TCM cells given IV
  Other Names: allogeneic CMV-specific CTLs

SUMMARY:
This phase I/II trial studies the safety and toxicity of post-transplant treatment with donor T cells engineered to express a chimeric antigen receptor (CAR) targeting CD19 in patients who have had a matched related allogeneic hematopoietic stem cell transplant for a CD19+ B cell malignancy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and feasibility of pre-emptive adoptive T cell therapy using ex vivo expanded cytomegalovirus (CMV)- or Epstein-Barr virus (EBV)-specific T cells derived from donor CD62L+ central memory (TCM) cells and genetically modified to express a CD19-specific chimeric antigen receptor (CAR) in patients in complete remission after human leukocyte antigen (HLA)-matched related donor hematopoietic stem cell transplantation (HCT) for CD19+ B cell malignancies at high risk of post-HCT relapse. (Cohort A)

II. To assess the safety and feasibility of adoptive T cell therapy using ex vivo expanded CMV- or EBV-specific T cells derived from donor CD62L+ TCM cells and genetically modified to express a CD19-specific CAR in patients with persistent, progressive or relapsed disease after HLA-matched related donor HCT for CD19+ B cell malignancies. (Cohort B)

SECONDARY OBJECTIVES:

I. To determine the duration of in vivo persistence of adoptively transferred bi-specific CD8+ T cells, and the phenotype of persisting T cells.

II. To determine if adoptively transferred bi-specific CD8+ T cells traffic to the bone marrow and function in vivo.

III. To determine if adoptively transferred bi-specific CD8+ T cells proliferate in allogeneic HCT recipients that reactivate CMV or EBV.

IV. To determine if the adoptive transfer of bi-specific CD8+ T cells eliminates CD19+ tumor cells in the subset of patients with a measurable tumor burden prior to T cell transfer.

OUTLINE:

At least 30 days after HCT, patients will receive one intravenous (IV) infusion of CMV/CD19 or EBV/CD19 bi-specific CD8+ T cells.

After completion of study treatment, patients are followed up periodically for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CD19+ B cell malignancy who have persistent, relapsed or progressive disease after hematopoietic stem cell transplant from an human leukocyte antigen (HLA)-matched related donor OR patients with CD19+ B cell malignancy who are planned for or have had a hematopoietic stem cell transplant from an HLA-matched related donor and are at risk of relapse after HCT defined by any one of the disease-specific criteria listed below:

  * Philadelphia chromosome negative acute lymphoblastic leukemia:

    * Beyond first complete remission (CR) at the time of pre-transplant evaluation
    * Required > 1 cycle of induction chemotherapy to achieve CR
    * First morphologic CR but with evidence of minimal residual disease by flow cytometry, conventional cytogenetics, fluorescence in situ hybridization (FISH) or polymerase chain reaction (PCR)
    * First CR with poor risk cytogenetics (t(4:11), t(8;14), hypodiploidy, near triploidy or > 5 cytogenetic abnormalities) at diagnosis
    * Planned for or have had a reduced intensity conditioned or non-myeloablative transplant
  * Philadelphia positive acute lymphoblastic leukemia

    * Not in CR at the time of pre-transplant evaluation
    * In CR with the following features:

      * Intolerant or unwilling to use a TKI after HCT
      * Current or previous detection of cytogenetic abnormalities in addition to t(9;22) by conventional karyotyping, FISH or molecular methods
  * Chronic lymphocytic leukemia, or low grade B cell lymphomas:

    * Failed or ineligible for prior immunochemotherapy that included a purine analog and anti-CD20 monoclonal antibody AND a lymph node >= 5 cm at the time of pre-transplant evaluation
  * Mantle cell lymphoma:

    * Failed or ineligible for autologous transplant AND a lymph node >= 2 cm at the time of pre-transplant evaluation
  * Diffuse large B cell lymphomas, large B cell transformation of an indolent lymphoma or other aggressive B cell lymphomas

    * Failed or ineligible for autologous transplant AND not in CR at the time of pre-transplant evaluation
* Confirmation of tumor diagnosis and expression of CD19 after review by University of Washington Medical Center (UWMC) or Seattle Cancer Care Alliance (SCCA) pathology services
* The patient has signed the informed consent form for this study
* DONOR: Genotypic or phenotypic HLA-identical family members
* DONOR: Express one or more of the following combinations of viral serostatus and HLA allele:

  * CMV seropositive and HLA-A*0101 positive
  * CMV seropositive and HLA-A*0201 positive
  * CMV seropositive and HLA-B*0702 positive
  * CMV seropositive and HLA-B*0801 positive
  * EBV seropositive and HLA-A*0201 positive
  * EBV seropositive and HLA-B*0801 positive
* DONOR: Hematocrit >= 35% at enrollment
* DONOR: Age >= 18 years
* DONOR: The donor has signed the informed consent form for the study

Exclusion Criteria:

* Known central nervous system (CNS) tumor (CNS2 or CNS3) that is refractory to intrathecal chemotherapy and/or cranio-spinal radiation; patients with a history of CNS disease that has been effectively treated to CNS1 or lower evidence of disease will be eligible
* Human immunodeficiency virus (HIV) seropositive
* Significant medical or psychological conditions that would make them unsuitable candidates for T cell therapy
* Fertile patients unwilling to use contraception during and for 12 months after protocol enrollment
* Pregnant or breast-feeding
* DONOR: G-CSF administered within one month prior to the blood draw for T cell collection
* DONOR: Unable for any reason to provide a 400 ml blood draw
* DONOR: Inadequate peripheral veins for blood collection
* DONOR: HIV-1, HIV-2, human T-lymphotropic virus (HTLV)-1 or HTLV-2 seropositive
* DONOR: Active hepatitis B or hepatitis C virus infection
* DONOR: Positive serologic test for syphilis
* DONOR: Aberrant CD45RA isoform expression on all T cells
* DONOR: Systolic blood pressure (BP) < 80 or > 200
* DONOR: Heart rate < 50 or > 120, if considered due to cardiac disease
* DONOR: Oxygen (O2) saturation < 88% on room air
* DONOR: Serum creatinine (Cr) > 3.0
* DONOR: Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 4 x the upper limit of normal
* DONOR: Unable to provide informed consent to participate
* DONOR: Significant medical conditions (e.g. immunosuppressive therapy) that would make them unsuitable T cell donors
* DONOR: Pregnant or nursing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity assessment of study treatment | Up to day 42 after the T cell infusion
  Incidence of grade >= 3 toxicity, as defined by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 occurring from the T cell infusion through day 42 after the T cell infusion. Analysis will be performed separately in patients in complete remission (cohort A) or with detectable disease (cohort B) at day 28 post-transplant (prior to the T cell infusion). Incidence of acute GVHD occurring from the T cell infusion through day 42 after the T cell infusion will be assessed.
Feasibility assessment of study treatment | Up to 5 years
  If the prescribed T cell dose is delivered in more than 50% of the patients, this approach will be considered feasible for further study to reduce relapse after allogeneic HCT.

SECONDARY OUTCOMES:
Anti-tumor efficacy and duration of persistence, migration, and function of adoptively transferred bi-specific effector cells | Up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Turtle, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338